CLINICAL TRIAL: NCT00550862
Title: A Study of INT 747 (6α-ethyl Chenodeoxycholic Acid (6-ECDCA)) in Combination With Ursodeoxycholic Acid (URSO®, UDCA) in Patients With Primary Biliary Cirrhosis
Brief Title: Study of INT 747 in Combination With URSO in Patients With Primay Biliary Cirrhosis (PBC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study stopped by sponsor due to administrative reasons
Sponsor: Intercept Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 747-202
Record Dates: First submitted 2007-10-27; First posted 2007-10-30 (Estimated); Results first posted 2012-01-23 (Estimated); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: Liver Cirrhosis, Biliary
Keywords: PBC, Primary Biliary Cirrhosis, Liver,
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — obeticholic acid; Ursodeoxycholic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- INT-747 10 mg (Experimental): INT-747 10 mg once daily in combination with URSO for 12 weeks.
  Interventions: Drug: INT-747; Drug: Ursodeoxycholic Acid (URSO)
- INT-747 25 mg (Experimental): INT-747 25 mg once daily in combination with URSO for 12 weeks.
  Interventions: Drug: INT-747; Drug: Ursodeoxycholic Acid (URSO)
- INT-747 50 mg (Experimental): INT-747 50 mg once daily in combination with URSO for 12 weeks.
  Interventions: Drug: INT-747; Drug: Ursodeoxycholic Acid (URSO)
- Placebo (Placebo Comparator): Placebo once daily in combination with URSO for 12 weeks.
  Interventions: Drug: INT-747; Drug: Ursodeoxycholic Acid (URSO); Drug: Placebo

INTERVENTIONS:
Drug: INT-747 — Once a day (QD) by mouth (PO)
  Other Names: Obeticholic acid (OCA), 6-ECDCA
Drug: Ursodeoxycholic Acid (URSO) — Stable dose for at least 6 months prior to screening. Dose as prescribed by physician.
  Other Names: URSO, UDCA
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The primary hypothesis is that INT-747 will cause a reduction in alkaline phosphatase levels in Primary Biliary Cirrhosis patients, over a 12 week treatment period, as compared to placebo.

DETAILED DESCRIPTION:
None provided

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 18 to 70 years.
* Stable dose of ursodeoxycholic acid (URSO, UDCA) for at least 6 months prior to screening.
* Female patients must be postmenopausal, surgically sterile, or prepared to use 2 methods of contraception with all sexual partners during the study and for 14 days after the end of dosing.
* Male patients must be prepared to use 2 methods of contraception with all sexual partners during the study and for 14 days after the end of the dosing.
* Proven or likely PBC, as demonstrated by the patient presenting with at least 2 of the following 3 diagnostic factors:

  1. History of increased AP levels for at least 6 months prior to Day 0
  2. Positive AMA titer (>1:40 titer on immunofluorescence or M2 positive by ELISA) or PBC-specific antinuclear antibodies (antinuclear dot and nuclear rim positive)
  3. Liver biopsy consistent with PBC.
* Screening AP value between 1.5 and 10 × ULN.

Exclusion Criteria:

* Administration of the following drugs at any time during the 3 months prior to screening for the study: colchicine, methotrexate, azathioprine, or systemic corticosteroids.
* Screening conjugated (direct) bilirubin >2 × ULN.
* Screening ALT or AST >5 × ULN.
* Screening serum creatinine >1.5 mg/dL (133 mol/L).
* History or presence of hepatic decompensation (e.g., variceal bleeds, encephalopathy, or poorly controlled ascites).
* History or presence of other concomitant liver diseases including hepatitis due to hepatitis B or C virus (HCV, HBV) infection, primary sclerosing cholangitis (PSC), alcoholic liver disease, definite autoimmune liver disease or biopsy proven nonalcoholic steatohepatitis (NASH).
* Pregnancy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2007-10 (Actual); Primary Completion 2009-08 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A Shapiro, MD, Study Director — Intercept Pharmaceuticals - Chief Medical Officer
Locations (32):
- United States (13):
  - U Florida Hepatology, Gainesville, Florida
  - University of Miami - Center for Liver Diseases, Miami, Florida
  - Tufts Medical Center, Boston, Massachusetts
  - Henry Ford Health Center Columbus, Novi, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Saint Louis University, St Louis, Missouri
  - Beth Israel Medical Center, New York, New York
  - Mt. Sinai School of Medicine, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - UT Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - McGuire DVAMC, Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
- Karls-Franzens University, Graz, Austria
- Canada (5):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - University of Manitoba, Winnipeg, Manitoba
  - University of Toronto Western Hospital, Toronto, Ontario
  - Centre de Recherche du CHUM / University of Montreal, Montreal, Quebec
- Hopital de l'Hotel Dieu, Lyon, France
- Germany (4):
  - Johann Wolfgang Goethe University, Frankfurt
  - University Medical Centre Hamburg-Eppendorf, Hamburg
  - Medical School of Hannover, Hanover
  - University of Munich, Munich
- Netherlands (2):
  - AMC University of Amsterdam, Amsterdam
  - Erasmus Medical Centre, Rotterdam
- Hospital Clinic i Provincial, Barcelona, Spain
- United Kingdom (5):
  - Queen Elizabeth Medical Center, Edgbaston, Birmingham
  - Royal Free Hospital, Hampstead, London
  - John Radcliffe Hospital, Headington, Oxford
  - Royal Infirmary, Edinburgh
  - University Upon Tyne/Newcastle, Newcastle upon Tyne

REFERENCES:
- [Derived] Hirschfield GM, Mason A, Luketic V, Lindor K, Gordon SC, Mayo M, Kowdley KV, Vincent C, Bodhenheimer HC Jr, Pares A, Trauner M, Marschall HU, Adorini L, Sciacca C, Beecher-Jones T, Castelloe E, Bohm O, Shapiro D. Efficacy of obeticholic acid in patients with primary biliary cirrhosis and inadequate response to ursodeoxycholic acid. Gastroenterology. 2015 Apr;148(4):751-61.e8. doi: 10.1053/j.gastro.2014.12.005. Epub 2014 Dec 11. PMID 25500425

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an international, multi-center, randomized, double-blind, placebo-controlled, multi-dose study with the majority of the sites being academic centers.
Pre-assignment Details: A total of 165 participants were enrolled into the double-blind phase of the study. Of these, 78 participants (21 of whom had received placebo) entered the open-label long-term safety extension (LTSE) phase
Groups:
- Obeticholic Acid (OCA) 10 Milligrams (mg): Participants were randomized to receive OCA 10 mg orally as a capsule once daily from Day 1 to Day 85 approximately 30 minutes before breakfast with water. Participants were instructed to swallow the capsule whole and not to chew, divide, or crush the capsule. Per the titration strategy, the participants were administered investigational product once every 3 days in the first week, once every 2 days in the second week, and daily from the third week onwards until end of study (EOS) (Day 85).
- OCA 25 mg: Participants were randomized to receive OCA 25 mg orally as a capsule once daily from Day 1 to Day 85 approximately 30 minutes before breakfast with water. Participants were instructed to swallow the capsule whole and not to chew, divide, or crush the capsule. Per the titration strategy, the participants were administered investigational product once every 3 days in the first week, once every 2 days in the second week, and daily from the third week onwards until EOS (Day 85).
- OCA 50 mg: Participants were randomized to receive OCA 50 mg orally as a capsule once daily from Day 1 to Day 85 approximately 30 minutes before breakfast with water. Participants were instructed to swallow the capsule whole and not to chew, divide, or crush the capsule. Per the titration strategy, the participants were administered investigational product once every 3 days in the first week, once every 2 days in the second week, and daily from the third week onwards until EOS (Day 85).
- Placebo: Participants were randomized to receive placebo orally as a capsule once daily from Day 1 to Day 85 approximately 30 minutes before breakfast with water. Participants were instructed to swallow the capsule whole and not to chew, divide, or crush the capsule. Per the titration strategy, the participants were administered investigational product once every 3 days in the first week, once every 2 days in the second week, and daily from the third week onwards until EOS (Day 85).
- LTSE OCA Total: A total of 78 participants from the double-blind phase entered the open-label LTSE phase of the study. Seven participants entered the LTSE within 2 weeks of completing the double-blind phase. Participants initially started dosing at less than or equal to (<=) 10 mg daily OCA and doses up to 50 mg daily were evaluated. Entry of 71 participants from double-blind phase to LTSE phase was delayed up to 10 months due to administrative reasons. All participants received open-label OCA during the LTSE phase of the study. Eligible participant who completed the DB phase were enrolled into the LTSE phase.
Period: Double-Blind Phase (Day 1 to Day 85)
Arm/Group | Obeticholic Acid (OCA) 10 Milligrams (mg) | OCA 25 mg | OCA 50 mg | Placebo | LTSE OCA Total
Started | 38 | 48 | 41 | 38 | 0
Completed | 32 | 42 | 25 | 37 | 0
Not Completed | 6 | 6 | 16 | 1 | 0
Not completed — Adverse Event | 5 | 5 | 12 | 1 | 0
Not completed — Elevated conjugated (direct) bilirubin | 1 | 0 | 2 | 0 | 0
Not completed — Elevated aspartate transaminase (AST)/ alanine transaminase (ALT) levels | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0
Period: LTSE Phase (Up to 12 Months)
Arm/Group | Obeticholic Acid (OCA) 10 Milligrams (mg) | OCA 25 mg | OCA 50 mg | Placebo | LTSE OCA Total
Started | 0 | 0 | 0 | 0 | 78
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 78
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 14
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 2
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 0 | 2
Not completed — Other: Study stopped by sponsor due to administrative reasons | 0 | 0 | 0 | 0 | 59

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Obeticholic Acid (OCA) 10 Milligrams (mg) | OCA 25 mg | OCA 50 mg | Placebo | Total
Number analyzed (Participants) | 38 | 48 | 41 | 38 | 165
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.6 (9.3) | 55.9 (8.0) | 54.0 (9.7) | 54.8 (8.5) | 55.1 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 45 | 38 | 36 | 157
  Male | 0 | 3 | 3 | 2 | 8
Race/Ethnicity, Customized [Number; unit: participants]
  White | 37 | 47 | 40 | 34 | 158
  Black | 0 | 0 | 1 | 1 | 2
  Asian | 1 | 0 | 0 | 1 | 2
  Other | 0 | 1 | 0 | 2 | 3
Region of Enrollment [Number; unit: participants]
  France | 1 | 1 | 0 | 0 | 2
  United States | 15 | 21 | 19 | 17 | 72
  Canada | 13 | 15 | 14 | 13 | 55
  Spain | 1 | 2 | 1 | 2 | 6
  Austria | 1 | 2 | 2 | 1 | 6
  Germany | 2 | 3 | 2 | 1 | 8
  Netherlands | 1 | 1 | 1 | 1 | 4
  United Kingdom | 4 | 3 | 2 | 3 | 12

OUTCOME MEASURES:

1. Primary Outcome: Double-blind Phase: Percent Change From Baseline in Serum Alkaline Phosphatase (ALP)
Description: Blood samples were collected for the analysis of serum ALP. Baseline was defined as the last observed value before the first dose of investigational product (Day 0). Percent change from Baseline was calculated as Post Baseline minus Baseline value divided by Baseline value and multiplied by 100.
Time Frame: Baseline and Up to Day 85
Population: Modified Intent-to-Treat (mITT) Population (N=161) comprised of all randomized participants who received at least 1 dose of investigational product and had at least 1 post-Baseline ALP evaluation taken ≤7 days after their last dose of investigational product.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Obeticholic Acid (OCA) 10 Milligrams (mg) | OCA 25 mg | OCA 50 mg | Placebo
Number analyzed (Participants) | 38 | 47 | 39 | 37
Percent change | -23.7 (17.8) | -24.7 (17.9) | -21.0 (27.6) | -2.6 (12.5)
Statistical Analysis 1: Comparison: Obeticholic Acid (OCA) 10 Milligrams (mg) vs Placebo; All tests: Descriptive methods were used with nominal p values provided and 95% confidence intervals; Test type: Other; p < 0.0001, Wilcoxon (Mann-Whitney) — Initial Phase 2 study: no a priori estimate of treatment effect available. Effect size estimated; Hierarchical model applied and pairwise comparisons of the 10mg treatment group versus the placebo group, then 25 mg and 50 mg were performed
Statistical Analysis 2: Comparison: OCA 25 mg vs Placebo; All tests: Descriptive methods were used with nominal p values provided and 95% confidence intervals; Test type: Other; p < 0.0001, Wilcoxon (Mann-Whitney) — Initial Phase 2 study: no a priori estimate of treatment effect available. Effect size estimated; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: OCA 50 mg vs Placebo; All tests: Descriptive methods were used with nominal p values provided and 95% confidence intervals; Test type: Other; p < 0.0001, Wilcoxon (Mann-Whitney) — Initial Phase 2 study: no a priori estimate of treatment effect available. Effect size estimated; [statistical method as in outcome 1, analysis 1]

2. Secondary Outcome: Double-blind Phase: Absolute Values for Serum ALP, Aspartate Aminotransferase (AST), Alanine Transaminase (ALT) and Gamma-glutamyl Transferase (GGT) Levels
Description: Blood samples were collected for the analysis of serum chemistry parameters including ALP, AST, ALT and GGT. Baseline was defined as the last observed value before the first dose of investigational product (Day 0).
Time Frame: Baseline and at Days 15, 29, 57 and 85
Population: Intent-to-Treat (ITT) Population (N=165) comprises all randomized participants who received at least 1 dose of investigational product. Only those participants with data available at specified timepoints has been presented.
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | Obeticholic Acid (OCA) 10 Milligrams (mg) | OCA 25 mg | OCA 50 mg | Placebo
Number analyzed (Participants) | 38 | 48 | 41 | 38
Units per liter
  ALP, Baseline | 294.4 (149.4) | 290.0 (123.6) | 289.5 (106.2) | 275.2 (102.7)
  ALP, Day 15: number analyzed (Participants) | 38 | 46 | 33 | 36
  ALP, Day 15 | 247.6 (117.9) | 239.3 (113.6) | 231.2 (87.5) | 269.2 (105.6)
  ALP, Day 29: number analyzed (Participants) | 35 | 43 | 27 | 37
  ALP, Day 29 | 227.2 (105.0) | 219.2 (100.5) | 216.1 (90.5) | 266.1 (118.0)
  ALP, Day 57: number analyzed (Participants) | 33 | 41 | 26 | 36
  ALP, Day 57 | 212.6 (98.9) | 231.7 (177.6) | 189.2 (67.5) | 271.5 (123.0)
  ALP, Day 85: number analyzed (Participants) | 38 | 48 | 40 | 38
  ALP, Day 85 | 219.0 (113.5) | 225.0 (169.1) | 227.9 (115.9) | 270.7 (118.7)
  AST, Baseline | 49 (22) | 44 (23) | 48 (24) | 42 (19)
  AST, Day 15: number analyzed (Participants) | 38 | 46 | 33 | 36
  AST, Day 15 | 44 (23) | 38 (19) | 47 (34) | 41 (17)
  AST, Day 29: number analyzed (Participants) | 35 | 43 | 27 | 37
  AST, Day 29 | 37 (13) | 36 (19) | 43 (28) | 42 (20)
  AST, Day 57: number analyzed (Participants) | 33 | 41 | 26 | 36
  AST, Day 57 | 36 (14) | 40 (45) | 37 (17) | 45 (28)
  AST, Day 85: number analyzed (Participants) | 38 | 48 | 40 | 38
  AST, Day 85 | 40 (23) | 37 (25) | 41 (24) | 41 (17)
  ALT, Baseline | 51 (29) | 51 (36) | 53 (35) | 47 (26)
  ALT, Day 15: number analyzed (Participants) | 38 | 46 | 33 | 36
  ALT, Day 15 | 40 (20) | 37 (28) | 49 (49) | 48 (24)
  ALT, Day 29: number analyzed (Participants) | 35 | 43 | 27 | 37
  ALT, Day 29 | 35 (15) | 32 (25) | 43 (40) | 46 (25)
  ALT, Day 57: number analyzed (Participants) | 33 | 41 | 26 | 36
  ALT, Day 57 | 32 (16) | 39 (70) | 34 (23) | 49 (29)
  ALT, Day 85: number analyzed (Participants) | 38 | 48 | 40 | 38
  ALT, Day 85 | 34 (20) | 34 (38) | 39 (32) | 45 (24)
  GGT, Baseline | 228 (212) | 273 (267) | 231 (182) | 189 (139)
  GGT, Day 15: number analyzed (Participants) | 38 | 46 | 33 | 36
  GGT, Day 15 | 137 (119) | 155 (197) | 108 (88) | 190 (141)
  GGT, Day 29: number analyzed (Participants) | 35 | 43 | 27 | 37
  GGT, Day 29 | 108 (92) | 109 (153) | 93 (90) | 196 (158)
  GGT, Day 57: number analyzed (Participants) | 33 | 41 | 26 | 36
  GGT, Day 57 | 96 (91) | 104 (189) | 76 (86) | 195 (165)
  GGT, Day 85: number analyzed (Participants) | 38 | 48 | 40 | 38
  GGT, Day 85 | 107 (124) | 115 (178) | 95 (89) | 209 (170)
Statistical Analysis 1: Comparison: Obeticholic Acid (OCA) 10 Milligrams (mg) vs OCA 25 mg vs OCA 50 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Double-blind Phase: Percent Change From Baseline in Serum ALP, AST, ALT and GGT Levels
Description: Blood samples were collected for the analysis of serum chemistry parameters including ALP, AST, ALT and GGT. Baseline was defined as the last observed value before the first dose of investigational product (Day 0). Percent change from Baseline was calculated as Post Baseline minus Baseline value divided by Baseline value and multiplied by 100.
Time Frame: Baseline and at Days 15, 29, 57 and 85
Population: ITT Population (N=165). Only those participants with data available at specified timepoints has been presented (n=164).
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Obeticholic Acid (OCA) 10 Milligrams (mg) | OCA 25 mg | OCA 50 mg | Placebo
Number analyzed (Participants) | 38 | 48 | 40 | 38
Percent change
  ALP, Day 15: number analyzed (Participants) | 38 | 46 | 33 | 36
  ALP, Day 15 | -13.5 (12.8) | -17.3 (9.8) | -16.1 (21.9) | -2.6 (10.8)
  ALP, Day 29: number analyzed (Participants) | 35 | 43 | 27 | 37
  ALP, Day 29 | -20.8 (14.2) | -23.4 (12.3) | -25.0 (17.5) | -4.6 (12.4)
  ALP, Day 57: number analyzed (Participants) | 33 | 41 | 26 | 36
  ALP, Day 57 | -26.0 (15.4) | -22.0 (17.2) | -29.0 (18.6) | -0.9 (17.1)
  ALP, Day 85 | -23.3 (17.1) | -24.0 (18.8) | -20.0 (27.4) | -2.6 (12.4)
  AST, Day 15: number analyzed (Participants) | 38 | 46 | 33 | 36
  AST, Day 15 | -6 (42) | -14 (18) | 13 (119) | 3 (23)
  AST, Day 29: number analyzed (Participants) | 35 | 43 | 27 | 37
  AST, Day 29 | -16 (22) | -17 (18) | -13 (26) | 2 (27)
  AST, Day 57: number analyzed (Participants) | 33 | 41 | 26 | 36
  AST, Day 57 | -19 (22) | -13 (30) | -15 (27) | 20 (95)
  AST, Day 85 | -17 (21) | -16 (20) | -9 (38) | -0 (23)
  ALT, Day 15: number analyzed (Participants) | 38 | 46 | 33 | 36
  ALT, Day 15 | -11 (61) | -26 (18) | 12 (176) | 6 (30)
  ALT, Day 29: number analyzed (Participants) | 35 | 43 | 27 | 37
  ALT, Day 29 | -25 (28) | -33 (18) | -29 (27) | 1 (31)
  ALT, Day 57: number analyzed (Participants) | 33 | 41 | 26 | 36
  ALT, Day 57 | -31 (23) | -32 (33) | -35 (24) | 8 (43)
  ALT, Day 85 | -28 (27) | -35 (22) | -21 (49) | -0 (35)
  GGT, Day 15: number analyzed (Participants) | 38 | 46 | 33 | 36
  GGT, Day 15 | -35 (14) | -43 (14) | -49 (12) | -1 (15)
  GGT, Day 29: number analyzed (Participants) | 35 | 43 | 27 | 37
  GGT, Day 29 | -48 (19) | -61 (15) | -63 (16) | 1 (24)
  GGT, Day 57: number analyzed (Participants) | 33 | 41 | 26 | 36
  GGT, Day 57 | -53 (26) | -64 (24) | -67 (18) | 2 (20)
  GGT, Day 85 | -48 (30) | -63 (24) | -57 (31) | 7 (28)
Statistical Analysis 1: Comparison: Obeticholic Acid (OCA) 10 Milligrams (mg) vs OCA 25 mg vs OCA 50 mg vs Placebo; Test type: Superiority or Other; p < 0.0005, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: LTSE Phase: Mean Percent Change From Baseline in Serum ALP, AST, ALT and GGT Levels
Description: Blood samples were collected for the analysis of serum chemistry parameters including ALP, AST, ALT and GGT. Baseline was defined as the last observed value before the first dose of investigational product (Day 85). Percent change from Baseline was calculated as Post Baseline minus Baseline value divided by Baseline value and multiplied by 100.
Time Frame: Baseline and at 3, 6, 9 and 12 Months
Population: Safety Population (N=78) comprised of all randomized participants who received at least 1 dose of investigational product. Only those participants with data available at specified timepoints has been presented (n=69).
Measure: Mean (Standard Deviation); unit: Percent change
Groups:
- LTSE OCA Total: A total of 78 participants from the double-blind phase entered the open-label LTSE phase of the study. Seven participants entered the LTSE within 2 weeks of completing the double-blind phase. Participants initially started dosing at less than or equal to (<=) 10 mg daily OCA and doses up to 50 mg daily were evaluated. Entry of 71 participants from double-blind phase to LTSE phase was delayed up to 10 months due to administrative reasons. All participants received open-label OCA during the LTSE phase of the study
Arm/Group | LTSE OCA Total
Number analyzed (Participants) | 69
Percent change
  ALP, 3-Month | -22.2 (18.2)
  ALP, 6-Month: number analyzed (Participants) | 68
  ALP, 6-Month | -23.7 (22.7)
  ALP, 9-Month: number analyzed (Participants) | 65
  ALP, 9-Month | -25.3 (22.2)
  ALP, 12-Month: number analyzed (Participants) | 61
  ALP, 12-Month | -26.5 (22.0)
  AST, 3-Month | 2.3 (29.2)
  AST, 6-Month: number analyzed (Participants) | 68
  AST, 6-Month | -1.2 (26.6)
  AST, 9-Month: number analyzed (Participants) | 65
  AST, 9-Month | -4.7 (27.1)
  AST, 12-Month: number analyzed (Participants) | 61
  AST, 12-Month | -0.7 (27.1)
  ALT, 3-Month | -17.8 (28.5)
  ALT, 6-Month: number analyzed (Participants) | 68
  ALT, 6-Month | -22.9 (26.5)
  ALT, 9-Month: number analyzed (Participants) | 65
  ALT, 9-Month | -23.3 (40.7)
  ALT, 12-Month: number analyzed (Participants) | 61
  ALT, 12-Month | -20.7 (26.4)
  GGT, 3-Month | -52.4 (25.4)
  GGT, 6-Month: number analyzed (Participants) | 68
  GGT, 6-Month | -57.5 (33.3)
  GGT, 9-Month: number analyzed (Participants) | 65
  GGT, 9-Month | -60.9 (24.9)
  GGT, 12-Month: number analyzed (Participants) | 61
  GGT, 12-Month | -60.4 (25.5)

5. Secondary Outcome: Double-blind Phase: Absolute Values for Albumin Levels
Description: Blood samples were collected for the analysis of serum chemistry parameter: Albumin. Baseline was defined as the last observed value before the first dose of investigational product (Day 0).
Time Frame: Baseline and at Days 15, 29, 57 and 85
Population: ITT Population (N=165). Only those participants with data available at specified timepoints has been presented.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Obeticholic Acid (OCA) 10 Milligrams (mg) | OCA 25 mg | OCA 50 mg | Placebo
Number analyzed (Participants) | 38 | 48 | 41 | 38
Grams per liter
  Baseline | 40.14 (4.66) | 41.17 (3.85) | 42.41 (2.77) | 42.03 (3.23)
  Day 15: number analyzed (Participants) | 38 | 46 | 33 | 36
  Day 15 | 39.84 (4.33) | 41.12 (3.59) | 41.15 (3.05) | 41.84 (3.38)
  Day 29: number analyzed (Participants) | 35 | 43 | 27 | 37
  Day 29 | 40.01 (3.38) | 40.94 (3.74) | 41.05 (3.64) | 41.21 (3.50)
  Day 57: number analyzed (Participants) | 33 | 42 | 26 | 36
  Day 57 | 40.29 (3.65) | 41.04 (3.90) | 41.76 (3.00) | 40.50 (4.33)
  Day 85 | 39.95 (4.19) | 41.09 (4.01) | 41.24 (3.86) | 41.69 (4.05)

6. Secondary Outcome: Double-blind Phase: Percent Change From Baseline in Albumin Levels
Description: Blood samples were collected for the analysis of serum chemistry parameter: Albumin. Baseline was defined as the last observed value before the first dose of investigational product (Day 0). Percent change from Baseline was calculated as Post Baseline minus Baseline value divided by Baseline value and multiplied by 100.
Time Frame: Baseline and at Days 15, 29, 57 and 85
Population: ITT Population (N=165). Only those participants with data available at specified timepoints has been presented.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Obeticholic Acid (OCA) 10 Milligrams (mg) | OCA 25 mg | OCA 50 mg | Placebo
Number analyzed (Participants) | 38 | 48 | 41 | 38
Percent change
  Day 15: number analyzed (Participants) | 38 | 46 | 33 | 36
  Day 15 | -0.42 (5.68) | -0.29 (5.71) | -2.66 (4.70) | -0.41 (5.18)
  Day 29: number analyzed (Participants) | 35 | 43 | 27 | 37
  Day 29 | -1.62 (4.52) | -0.73 (5.10) | -2.59 (5.69) | -1.97 (4.78)
  Day 57: number analyzed (Participants) | 33 | 42 | 26 | 36
  Day 57 | -0.69 (5.56) | -0.26 (4.83) | -2.00 (4.27) | -3.58 (6.90)
  Day 85 | -0.13 (5.03) | -0.11 (5.42) | -2.82 (6.04) | -0.82 (5.79)

7. Secondary Outcome: Double-blind Phase: Absolute Values for Conjugated (Direct) Bilirubin
Description: Blood samples were collected for the analysis of serum chemistry parameter: Conjugated (Direct) bilirubin. Baseline was defined as the last observed value before the first dose of investigational product (Day 0).
Time Frame: Baseline and at Days 15, 29, 57 and 85
Population: ITT Population (N=165). Only those participants with data available at specified timepoints has been presented.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Obeticholic Acid (OCA) 10 Milligrams (mg) | OCA 25 mg | OCA 50 mg | Placebo
Number analyzed (Participants) | 38 | 48 | 41 | 38
Micromoles per liter
  Baseline | 4.2 (3.1) | 3.9 (2.4) | 4.7 (3.3) | 3.6 (2.8)
  Day 15: number analyzed (Participants) | 38 | 46 | 33 | 36
  Day 15 | 4.9 (5.0) | 3.1 (2.2) | 3.3 (2.2) | 3.4 (2.4)
  Day 29: number analyzed (Participants) | 34 | 43 | 27 | 37
  Day 29 | 3.3 (2.6) | 3.3 (2.6) | 5.6 (14.4) | 3.7 (2.8)
  Day 57: number analyzed (Participants) | 33 | 41 | 26 | 36
  Day 57 | 3.4 (3.1) | 3.4 (2.6) | 3.0 (1.6) | 3.5 (3.0)
  Day 85: number analyzed (Participants) | 38 | 48 | 40 | 38
  Day 85 | 3.9 (3.8) | 3.2 (2.7) | 5.5 (8.5) | 3.6 (3.2)

8. Secondary Outcome: Double-blind Phase: Percent Change From Baseline in Conjugated (Direct) Bilirubin
Description: Blood samples were collected for the analysis of serum chemistry parameter: Direct bilirubin. Baseline was defined as the last observed value before the first dose of investigational product (Day 0). Percent change from Baseline was calculated as Post Baseline minus Baseline value divided by Baseline value and multiplied by 100.
Time Frame: Baseline and at Days 15, 29, 57 and 85
Population: ITT Population (N=165). Only those participants with data available at specified timepoints has been presented (n=164).
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Obeticholic Acid (OCA) 10 Milligrams (mg) | OCA 25 mg | OCA 50 mg | Placebo
Number analyzed (Participants) | 38 | 48 | 40 | 38
Percent change
  Day 15: number analyzed (Participants) | 38 | 46 | 33 | 36
  Day 15 | 14.6 (60.9) | -15.3 (38.1) | -17.6 (35.4) | 2.7 (38.2)
  Day 29: number analyzed (Participants) | 34 | 43 | 27 | 37
  Day 29 | -3.3 (41.2) | -11.8 (43.7) | 31.3 (276.8) | 12.2 (39.3)
  Day 57: number analyzed (Participants) | 33 | 41 | 26 | 36
  Day 57 | -2.9 (39.6) | -8.8 (44.1) | -18.7 (31.3) | 1.4 (32.8)
  Day 85 | 0.0 (49.6) | -12.2 (40.0) | 10.0 (143.2) | 3.7 (48.2)

9. Secondary Outcome: LTSE Phase: Mean Percent Change From Baseline in Total and Conjugated (Direct) Bilirubin
Description: Blood samples were collected for the analysis of serum chemistry parameters Total and direct bilirubin. Baseline was defined as the last observed value before the first dose of investigational product (Day 85). Percent change from Baseline was calculated as Post Baseline minus Baseline value divided by Baseline value and multiplied by 100.
Time Frame: Baseline and at 3, 6, 9 and 12 Months
Population: Safety Population (N=78). Only those participants with data available at specified timepoints has been presented (n=69)
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | LTSE OCA Total
Number analyzed (Participants) | 69
Percent change
  Direct bilirubin, 3-Month | 19.6 (46.2)
  Direct bilirubin, 6-Month: number analyzed (Participants) | 68
  Direct bilirubin, 6-Month | 24.6 (53.2)
  Direct bilirubin, 9-Month: number analyzed (Participants) | 65
  Direct bilirubin, 9-Month | 15.2 (44.3)
  Direct bilirubin, 12-Month: number analyzed (Participants) | 61
  Direct bilirubin, 12-Month | 23.1 (68.3)
  Total bilirubin, 3-Month | -17.0 (28.0)
  Total bilirubin, 6-Month: number analyzed (Participants) | 68
  Total bilirubin, 6-Month | -11.6 (25.2)
  Total bilirubin, 9-Month: number analyzed (Participants) | 65
  Total bilirubin, 9-Month | -18.3 (29.7)
  Total bilirubin, 12-Month: number analyzed (Participants) | 61
  Total bilirubin, 12-Month | -8.9 (35.8)

10. Secondary Outcome: Double-blind Phase: Change From Baseline in Enhanced Liver Fibrosis (ELF) Score
Description: Enhanced Liver Fibrosis (ELF) combines measurements of tissue inhibitor of metalloprotein-ases-1 (TIMP-1), amino-terminal pro-peptide of type III procollagen (PIIINP), and hyaluronic acid (HA). The ELF score is calculated as: 2.278 + 0.851 ln (HA) + 0.751 ln (PIIINP) + 0.394 ln (TIMP-1). An ELF score of less than 7.7 indicates no to mild fibrosis; ≥ 7.7 - < 9.8: Moderate fibrosis; ≥ 9.8 - < 11.3: Severe fibrosis; ≥ 11.3: Cirrhosis. A negative change from Baseline indicates decreased fibrosis. Higher the ELF is associated with higher fibrosis stages and greater the risk of progression. A minimum and maximum value for the scale range does not exist for this assessment. Baseline was defined as the last observed value before the first dose of investigational product (Day 0). Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and up to Day 85
Population: ITT Population (N=165). Only those participants with data available at specified timepoints has been presented (n=146).
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Obeticholic Acid (OCA) 10 Milligrams (mg) | OCA 25 mg | OCA 50 mg | Placebo
Number analyzed (Participants) | 32 | 42 | 36 | 36
Scores on a scale | -0.095 (0.593) | 0.008 (0.561) | 0.124 (0.685) | -0.212 (0.627)

11. Secondary Outcome: Double-blind Phase: Change From Baseline in HA, P3NP, and TIMP-1 Levels
Description: Blood samples were collected for the analysis of extracellular matrix markers, including TIMP-1, PIIINP, and HA. The ELF score has been reported to show good correlations with fibrosis stages in chronic liver disease, with higher ELF scores associated with higher fibrosis stages. Baseline was defined as the last observed value before the first dose of investigational product (Day 0). Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and Up to Day 85
Population: ITT Population (N=165). Only those participants with data available at specified timepoints has been presented (n=146).
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Obeticholic Acid (OCA) 10 Milligrams (mg) | OCA 25 mg | OCA 50 mg | Placebo
Number analyzed (Participants) | 32 | 42 | 36 | 36
Nanograms per milliliter
  HA | -6.771 (59.677) | 12.287 (73.090) | 20.117 (97.056) | -21.359 (69.389)
  P3NP | -0.503 (3.017) | -0.468 (2.389) | 1.858 (6.547) | -0.943 (3.206)
  TIMP-1 | 15.341 (218.71) | -18.409 (191.768) | 43.921 (222.930) | -65.196 (257.295)

12. Secondary Outcome: Double-blind Phase: Absolute Values for Biomarkers of Hepatic Inflammation: C-reactive Protein
Description: Blood samples were collected for the analysis of biomarkers of hepatic inflammation including C-reactive protein. Baseline was defined as the last observed value before the first dose of investigational product (Day 0).
Time Frame: Baseline and Up to Day 85
Population: ITT Population (N=165). Only those participants with data available at specified timepoints has been presented (n-144).
Measure: Mean (Standard Deviation); unit: Milligrams per milliliter
Arm/Group | Obeticholic Acid (OCA) 10 Milligrams (mg) | OCA 25 mg | OCA 50 mg | Placebo
Number analyzed (Participants) | 36 | 41 | 35 | 32
Milligrams per milliliter
  Baseline | 7.9 (7.5) | 7.8 (8.9) | 5.2 (5.6) | 5.1 (4.6)
  Day 85: number analyzed (Participants) | 28 | 36 | 30 | 31
  Day 85 | 6.4 (7.2) | 4.0 (4.4) | 6.0 (13.2) | 6.0 (5.8)

13. Secondary Outcome: Double-blind Phase: Change From Baseline Values for Biomarkers of Hepatic Inflammation: C-reactive Protein
Description: Blood samples were collected for the analysis of biomarkers of hepatic inflammation including C-reactive protein. Baseline was defined as the last observed value before the first dose of investigational product (Day 0). Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and Up to Day 85
Population: ITT Population (N=165). Only those participants with data available at specified time points has been presented (n=114).
Measure: Mean (Standard Deviation); unit: Milligrams per milliliter
Arm/Group | Obeticholic Acid (OCA) 10 Milligrams (mg) | OCA 25 mg | OCA 50 mg | Placebo
Number analyzed (Participants) | 28 | 31 | 27 | 28
Milligrams per milliliter | -1.8 (7.9) | -3.7 (6.6) | 1.4 (9.4) | 0.3 (3.7)

14. Secondary Outcome: Double-blind Phase: Absolute Values for Biomarkers of Hepatic Inflammation: Non-essential Fatty Acid (NEFA)
Description: Blood samples were collected for the analysis of biomarkers of hepatic inflammation including NEFA. Baseline was defined as the last observed value before the first dose of investigational product (Day 0).
Time Frame: Baseline and Up to Day 85
Population: ITT Population (N=165). Only those participants with data available at specified timepoints has been presented (n=143).
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Obeticholic Acid (OCA) 10 Milligrams (mg) | OCA 25 mg | OCA 50 mg | Placebo
Number analyzed (Participants) | 35 | 41 | 35 | 32
Millimoles per liter
  Baseline | 0.58 (0.23) | 0.55 (0.24) | 0.62 (0.23) | 0.54 (0.26)
  Day 85: number analyzed (Participants) | 28 | 34 | 30 | 31
  Day 85 | 0.49 (0.24) | 0.51 (0.19) | 0.55 (0.25) | 0.56 (0.19)

15. Secondary Outcome: Double-blind Phase: Change From Baseline Values for Biomarkers of Hepatic Inflammation: NEFA
Description: Blood samples were collected for the analysis of biomarkers of hepatic inflammation including NEFA. Baseline was defined as the last observed value before the first dose of investigational product (Day 0). Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and Up to Day 85
Population: ITT Population (N=165). Only those participants with data available at specified time points has been presented (n=112).
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Obeticholic Acid (OCA) 10 Milligrams (mg) | OCA 25 mg | OCA 50 mg | Placebo
Number analyzed (Participants) | 27 | 30 | 27 | 28
Millimoles per liter | -0.06 (0.19) | -0.01 (0.27) | -0.07 (0.20) | 0.04 (0.25)

16. Secondary Outcome: Double-blind Phase: Absolute Values for Biomarkers of Hepatic Inflammation: Tumor Necrosis Factor Alpha (TNF-alpha)
Description: Blood samples were collected for the analysis of biomarkers of hepatic inflammation including TNF-alpha. Baseline was defined as the last observed value before the first dose of investigational product (Day 0).
Time Frame: Baseline and Up to Day 85
Population: ITT Population (N=165). Only those participants with data available at specified timepoints has been presented (n=144).
Measure: Mean (Standard Deviation); unit: Nanograms per liter
Arm/Group | Obeticholic Acid (OCA) 10 Milligrams (mg) | OCA 25 mg | OCA 50 mg | Placebo
Number analyzed (Participants) | 35 | 41 | 35 | 33
Nanograms per liter
  Baseline: number analyzed (Participants) | 35 | 41 | 35 | 32
  Baseline | 15.6 (7.1) | 13.8 (4.4) | 16.1 (11.7) | 11.4 (3.2)
  Day 85: number analyzed (Participants) | 29 | 38 | 31 | 33
  Day 85 | 18.1 (14.8) | 15.4 (7.3) | 16.2 (12.1) | 13.6 (4.5)

17. Secondary Outcome: Double-blind Phase: Change From Baseline Values for Biomarkers of Hepatic Inflammation: TNF-alpha
Description: Blood samples were collected for the analysis of biomarkers of hepatic inflammation including TNF-alpha. Baseline was defined as the last observed value before the first dose of investigational product (Day 0). Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and Up to Day 85
Population: ITT Population (N=165). Only those participants with data available at specified timepoints has been presented (n=119).
Measure: Mean (Standard Deviation); unit: Nanograms per liter
Arm/Group | Obeticholic Acid (OCA) 10 Milligrams (mg) | OCA 25 mg | OCA 50 mg | Placebo
Number analyzed (Participants) | 28 | 33 | 28 | 30
Nanograms per liter | 3.0 (15.6) | 1.7 (5.7) | -0.2 (15.8) | 1.2 (4.2)

18. Secondary Outcome: Double-blind Phase: Absolute Values for Biomarkers of Hepatic Inflammation: TNF-beta and Tumor Growth Factor Beta (TGF-beta)
Description: Blood samples were collected for the analysis of biomarkers of hepatic inflammation including TNF-beta and TGF-beta. Baseline was defined as the last observed value before the first dose of investigational product (Day 0).
Time Frame: Baseline and Up to Day 85
Population: ITT Population (N-165). Only those participants with data available at specified timepoints has been presented (142).
Measure: Mean (Standard Deviation); unit: Picomoles per liter
Arm/Group | Obeticholic Acid (OCA) 10 Milligrams (mg) | OCA 25 mg | OCA 50 mg | Placebo
Number analyzed (Participants) | 31 | 43 | 34 | 34
Picomoles per liter
  TNF-beta, Baseline: number analyzed (Participants) | 17 | 20 | 21 | 18
  TNF-beta, Baseline | 13.1 (14.8) | 10.8 (12.2) | 8.7 (10.4) | 8.8 (12.0)
  TNF-beta, Day 85: number analyzed (Participants) | 7 | 10 | 8 | 11
  TNF-beta, Day 85 | 11.0 (7.8) | 14.5 (17.0) | 6.7 (7.6) | 10.9 (17.3)
  TGF-beta, Baseline: number analyzed (Participants) | 31 | 39 | 34 | 29
  TGF-beta, Baseline | 35.6 (22.0) | 37.0 (23.3) | 26.2 (22.9) | 36.4 (25.3)
  TGF-beta, Day 85: number analyzed (Participants) | 30 | 43 | 34 | 34
  TGF-beta, Day 85 | 39.2 (22.9) | 41.0 (25.7) | 40.4 (22.3) | 30.1 (23.1)

19. Secondary Outcome: Double-blind Phase: Change From Baseline Values for Biomarkers of Hepatic Inflammation: TNF-beta and TGF-beta
Description: Blood samples were collected for the analysis of biomarkers of hepatic inflammation including TNF-beta and TGF-beta. Baseline was defined as the last observed value before the first dose of investigational product (Day 0). Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and Up to Day 85
Population: ITT Population (N=165). Only those participants with data available at specified time points has been presented (n=120).
Measure: Mean (Standard Deviation); unit: Picomoles per liter
Arm/Group | Obeticholic Acid (OCA) 10 Milligrams (mg) | OCA 25 mg | OCA 50 mg | Placebo
Number analyzed (Participants) | 26 | 35 | 31 | 28
Picomoles per liter
  TNF-beta: number analyzed (Participants) | 6 | 7 | 6 | 9
  TNF-beta | -11.3 (25.1) | 3.9 (6.1) | 2.2 (7.1) | 1.1 (11.2)
  TGF-beta | 3.7 (22.1) | 3.4 (27.9) | 14.0 (27.8) | 0.1 (30.0)

20. Secondary Outcome: Double-blind Phase: Absolute Values for Biomarkers of Hepatic Inflammation: Bile Acids and Glutathion
Description: Blood samples were collected for the analysis of biomarkers of hepatic inflammation including Bile acids and glutathion. Baseline was defined as the last observed value before the first dose of investigational product (Day 0).
Time Frame: Baseline and Up to Day 85
Population: ITT Population (N=165). Only those participants with data available at specified timepoints has been presented (n=144).
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Obeticholic Acid (OCA) 10 Milligrams (mg) | OCA 25 mg | OCA 50 mg | Placebo
Number analyzed (Participants) | 35 | 41 | 35 | 33
Micromoles per liter
  Bile acids, Baseline: number analyzed (Participants) | 34 | 41 | 35 | 32
  Bile acids, Baseline | 36.9 (31.7) | 29.5 (26.1) | 36.0 (48.9) | 27.6 (32.3)
  Bile acids, Day 85: number analyzed (Participants) | 29 | 37 | 31 | 33
  Bile acids, Day 85 | 37.8 (47.3) | 30.2 (42.9) | 34.6 (57.2) | 26.2 (29.2)
  Glutathione, Baseline: number analyzed (Participants) | 35 | 41 | 35 | 32
  Glutathione, Baseline | 3.7 (1.3) | 4.0 (1.9) | 3.4 (1.6) | 3.8 (1.8)
  Glutathione, Day 85: number analyzed (Participants) | 29 | 38 | 31 | 32
  Glutathione, Day 85 | 5.0 (2.1) | 5.3 (1.9) | 4.8 (2.0) | 4.8 (1.9)

21. Secondary Outcome: Double-blind Phase: Change From Baseline Values for Biomarkers of Hepatic Inflammation: Bile Acids and Glutathion
Description: Blood samples were collected for the analysis of biomarkers of hepatic inflammation including Bile acids and glutathion. Baseline was defined as the last observed value before the first dose of investigational product (Day 0). Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and Up to Day 85
Population: ITT Population (N=165). Only those participants with data available at specified time points has been presented (n=119).
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Obeticholic Acid (OCA) 10 Milligrams (mg) | OCA 25 mg | OCA 50 mg | Placebo
Number analyzed (Participants) | 28 | 33 | 28 | 30
Micromoles per liter
  Bile acids: number analyzed (Participants) | 27 | 32 | 28 | 30
  Bile acids | -1.4 (38.7) | -1.1 (36.3) | 0.5 (77.9) | -1.0 (28.3)
  Glutathione | 1.4 (1.7) | 1.3 (1.9) | 1.2 (1.4) | 1.0 (2.3)

22. Secondary Outcome: Double-blind Phase: Absolute Values for Biomarkers of Hepatic Inflammation: Immunoglobulin M (IgM)
Description: Blood samples were collected for the analysis of biomarkers of hepatic inflammation including IgM. Baseline was defined as the last observed value before the first dose of investigational product (Day 0).
Time Frame: Baseline and Up to Day 85
Population: ITT Population (N=165). Only those participants with data available at specified timepoints has been presented (n=144).
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Obeticholic Acid (OCA) 10 Milligrams (mg) | OCA 25 mg | OCA 50 mg | Placebo
Number analyzed (Participants) | 35 | 41 | 35 | 33
Grams per liter
  Baseline: number analyzed (Participants) | 35 | 41 | 35 | 32
  Baseline | 4.31 (2.12) | 3.13 (1.95) | 3.82 (3.35) | 3.06 (1.73)
  Day 85: number analyzed (Participants) | 29 | 38 | 31 | 33
  Day 85 | 3.73 (1.91) | 2.62 (1.76) | 3.02 (2.14) | 2.97 (1.61)

23. Secondary Outcome: Double-blind Phase: Change From Baseline Values for Biomarkers of Hepatic Inflammation: IgM
Description: Blood samples were collected for the analysis of biomarkers of hepatic inflammation including IgM. Baseline was defined as the last observed value before the first dose of investigational product (Day 0). Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and Up to Day 85
Population: ITT Population (N=165). Only those participants with data available at specified time points has been presented (n=119).
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Obeticholic Acid (OCA) 10 Milligrams (mg) | OCA 25 mg | OCA 50 mg | Placebo
Number analyzed (Participants) | 28 | 33 | 28 | 30
Grams per liter | -0.71 (0.94) | -0.58 (0.75) | -0.95 (1.57) | 0.02 (0.61)

24. Secondary Outcome: Double-blind Phase: Absolute Values for Biomarkers of Hepatic Inflammation: Osteopontin
Description: Blood samples were collected for the analysis of biomarkers of hepatic inflammation including Osteopontin. Baseline was defined as the last observed value before the first dose of investigational product (Day 0).
Time Frame: Baseline and Up to Day 85
Population: ITT Population (165). Only those participants with data available at specified timepoints has been presented (n=144).
Measure: Mean (Standard Deviation); unit: Micrograms per liter
Arm/Group | Obeticholic Acid (OCA) 10 Milligrams (mg) | OCA 25 mg | OCA 50 mg | Placebo
Number analyzed (Participants) | 35 | 41 | 35 | 33
Micrograms per liter
  Baseline | 305 (175) | 279 (118) | 286 (122) | 264 (130)
  Day 85: number analyzed (Participants) | 29 | 38 | 31 | 32
  Day 85 | 335 (187) | 318 (131) | 350 (170) | 245 (115)

25. Secondary Outcome: Double-blind Phase: Change From Baseline Values for Biomarkers of Hepatic Inflammation: Osteopontin
Description: Blood samples were collected for the analysis of biomarkers of hepatic inflammation including Osteopontin. Baseline was defined as the last observed value before the first dose of investigational product (Day 0). Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and Up to Day 85
Population: ITT Population (165). Only those participants with data available at specified time points has been presented (n=119).
Measure: Mean (Standard Deviation); unit: Micrograms per liter
Arm/Group | Obeticholic Acid (OCA) 10 Milligrams (mg) | OCA 25 mg | OCA 50 mg | Placebo
Number analyzed (Participants) | 28 | 33 | 28 | 30
Micrograms per liter | 51 (130) | 36 (141) | 72 (83) | -18 (119)

26. Secondary Outcome: Double-blind Phase: Absolute Values for Total Endogenous Bile Acids
Description: Serum samples were collected for the analysis total endogenous bile acids. Baseline was defined as the last observed value before the first dose of investigational product (Day 0).
Time Frame: Baseline and Up to Day 85
Population: ITT Population (N=165). Only those participants with data available at specified time points has been presented (n=143).
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Obeticholic Acid (OCA) 10 Milligrams (mg) | OCA 25 mg | OCA 50 mg | Placebo
Number analyzed (Participants) | 32 | 42 | 34 | 35
Micromoles per liter
  Baseline: number analyzed (Participants) | 32 | 42 | 34 | 32
  Baseline | 11.011 (9.071) | 10.013 (12.860) | 16.048 (28.325) | 6.350 (9.524)
  Day 85: number analyzed (Participants) | 29 | 40 | 33 | 35
  Day 85 | 9.516 (14.945) | 5.948 (15.590) | 23.935 (54.351) | 8.796 (11.557)

27. Secondary Outcome: Double-blind Phase: Change From Baseline in Total Endogenous Bile Acids
Description: Serum samples were collected for the analysis of total endogenous bile acids. Baseline was defined as the last observed value before the first dose of investigational product (Day 0). Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and Up to Day 85
Population: ITT Population (N=165). Only those participants with data available at specified time points has been presented (n=121).
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Obeticholic Acid (OCA) 10 Milligrams (mg) | OCA 25 mg | OCA 50 mg | Placebo
Number analyzed (Participants) | 25 | 38 | 29 | 29
Micromoles per liter | -4.489 (34.302) | -3.018 (29.937) | 33.526 (153.176) | 0.525 (19.238)

28. Secondary Outcome: Double-blind Phase: Absolute Values for Fibroblast Growth Factor 19 (FGF19)
Description: FGF-19 is a protein secreted by the gastro-intestine under farnesoid X receptor (FXR) control. Baseline was defined as the last observed value before the first dose of investigational product (Day 0).
Time Frame: Baseline and Up to Day 85
Population: ITT Population (N=165). Only those participants with data available at specified time points has been presented (n=143).
Measure: Mean (Standard Deviation); unit: Nanograms per liter
Arm/Group | Obeticholic Acid (OCA) 10 Milligrams (mg) | OCA 25 mg | OCA 50 mg | Placebo
Number analyzed (Participants) | 32 | 42 | 34 | 35
Nanograms per liter
  Baseline: number analyzed (Participants) | 32 | 42 | 34 | 32
  Baseline | 102.9 (60.7) | 104.1 (64.5) | 115.7 (122.4) | 84.1 (56.1)
  Day 85: number analyzed (Participants) | 29 | 40 | 33 | 35
  Day 85 | 248.2 (221.3) | 386.9 (443.9) | 2269.7 (9874.8) | 95.6 (65.6)

29. Secondary Outcome: Double-blind Phase: Percent Change From Baseline Values for FGF19
Description: FGF-19 is a protein secreted by the gastro-intestine under FXR control. Baseline was defined as the last observed value before the first dose of investigational product (Day 0). Percent change from Baseline was calculated as Post Baseline minus Baseline value divided by Baseline value and multiplied by 100.
Time Frame: Baseline and Up to Day 85
Population: ITT Population (N=165). Only those participants with data available at specified time points has been presented (n=126).
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Obeticholic Acid (OCA) 10 Milligrams (mg) | OCA 25 mg | OCA 50 mg | Placebo
Number analyzed (Participants) | 28 | 38 | 30 | 30
Percent change | 161.0 (148.7) | 464.7 (1419.1) | 3029.2 (13234.0) | 75.9 (250.6)

30. Secondary Outcome: Double-blind Phase: Change From Baseline to Day 85 in Quality of Life as Determined by Short Form-36 (SF-36) Scale
Description: The SF-36 determines participants' overall quality of life by assessing 1) limitations in physical functioning due to health problems; 2) limitations in usual role because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality; 6) limitations in social functioning because of physical or emotional problems; 7) limitations in usual role due to emotional problems; and 8) general mental health. Items 1-4 primarily contribute to the physical component summary (PCS) score of the SF-36. Items 5-8 primarily contribute to the mental component summary (MCS) score of the SF-36. These eight dimensions can be summarized numerically into two scores: PCS and MCS; with score range from 0=worst to 100=best, with higher scores indicating better health. Increases from baseline indicate improvement. Baseline was defined as Day 0. Change from Baseline was defined as value of post Baseline minus Baseline value.
Time Frame: Baseline and Up to Day 85
Population: ITT Population (N=165). Only those participants with data available at specified time points has been presented (n=153).
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Obeticholic Acid (OCA) 10 Milligrams (mg) | OCA 25 mg | OCA 50 mg | Placebo
Number analyzed (Participants) | 37 | 44 | 36 | 36
Scores on a scale
  PCS | -0.0 (5.5) | 0.1 (5.7) | 1.3 (7.3) | 1.1 (5.7)
  MCS | -2.2 (7.0) | -1.5 (4.8) | -1.2 (10.0) | 1.7 (9.3)

31. Secondary Outcome: LTSE Phase: Absolute Values of Quality of Life as Determined by SF-36 Scale
Description: The SF-36 determines participants' overall quality of life by assessing 1) limitations in physical functioning due to health problems; 2) limitations in usual role because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality; 6) limitations in social functioning because of physical or emotional problems; 7) limitations in usual role due to emotional problems; and 8) general mental health. Items 1-4 primarily contribute to the physical component summary (PCS) score of the SF-36. Items 5-8 primarily contribute to the mental component summary (MCS) score of the SF-36. These eight dimensions can be summarized numerically into two scores: PCS and MCS; with score range from 0=worst to 100=best, with higher scores indicating better health. Increases from baseline indicate improvement. Baseline was defined as Day 85
Time Frame: Baseline and at 3, 6, 9 and 12 Months
Population: ITT Population.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | LTSE OCA Total
Number analyzed (Participants) | 78
Scores on a scale
  Baseline, PCS | 45.7 (10.7)
  12 Months, PCS | 44.1 (11.2)
  Baseline, MCS | 49.4 (10.2)
  12 Months, MCS | 48.3 (11.2)

32. Secondary Outcome: Double-blind Phase: Change From Baseline in Quality of Life (QoL) as Determined by Primary Biliary Cirrhosis 40 (PBC-40) Scale
Description: PBC-40 is a disease-specific quality of life questionnaire,which consists of 5 Domains(score ranges):general symptoms (score range 7-35), itch (3-15), fatigue (11-55), cognitive function (6-30) and emotional (1-15); higher scores indicated worse outcomes.The 40 questions from the PBC-40 questionnaire were scored from 1 (lowest impact of PBC on QoL) to 5 (representing highest impact); Higher scores indicate worse quality of life. Outcomes of 'never', 'not at all' or 'strongly agree' are scored with 1, 'always', 'very much' or 'strongly disagree' with 5, with following exceptions: For questions 34-39 outcomes were scored in reverse,i.e., 'strongly agree' with 5, and 'strongly disagree' with 1. If less than 50% of the questions per domain were not answered, missing values were imputed by mean of the available question scores for that domain.If for any item multiple answers are given, most severe was used. Baseline = Day 0. Change from Baseline=post Baseline minus Baseline value.
Time Frame: Baseline and at Days 29, 57 and 85
Population: Safety Population. Only those participants with data available at specified time points has been presented (n=163).
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Obeticholic Acid (OCA) 10 Milligrams (mg) | OCA 25 mg | OCA 50 mg | Placebo
Number analyzed (Participants) | 38 | 47 | 40 | 38
Scores on a scale
  General symptoms, Day 29: number analyzed (Participants) | 35 | 44 | 28 | 36
  General symptoms, Day 29 | -0.4 (2.4) | -0.9 (2.5) | 0.3 (2.1) | -0.4 (1.9)
  General symptoms, Day 57: number analyzed (Participants) | 33 | 43 | 25 | 37
  General symptoms, Day 57 | 0.1 (2.7) | -0.5 (2.2) | 0.2 (1.9) | -0.3 (2.3)
  General symptoms, Day 85 | 0.3 (2.9) | 0.0 (2.8) | -0.1 (2.8) | -0.4 (2.2)
  Itch, Day 29: number analyzed (Participants) | 35 | 44 | 28 | 36
  Itch, Day 29 | 0.6 (2.2) | 2.0 (2.9) | 3.4 (3.7) | -0.2 (1.7)
  Itch, Day 57: number analyzed (Participants) | 33 | 43 | 25 | 37
  Itch, Day 57 | 0.6 (2.7) | 2.0 (3.0) | 2.9 (2.9) | -0.9 (1.7)
  Itch, Day 85 | 1.1 (2.6) | 1.6 (2.6) | 2.9 (3.2) | -0.8 (2.3)
  Fatigue, Day 29: number analyzed (Participants) | 35 | 44 | 28 | 37
  Fatigue, Day 29 | -0.5 (4.6) | -1.3 (5.1) | -0.8 (5.2) | -2.6 (4.2)
  Fatigue, Day 57: number analyzed (Participants) | 33 | 43 | 26 | 37
  Fatigue, Day 57 | -0.3 (4.7) | -0.6 (5.0) | -1.3 (5.3) | -3.5 (6.3)
  Fatigue, Day 85 | -0.4 (4.3) | 0.4 (4.6) | -0.3 (5.3) | -3.1 (4.6)
  Cognitive function, Day 29: number analyzed (Participants) | 35 | 44 | 28 | 37
  Cognitive function, Day 29 | -0.1 (2.0) | -0.5 (2.0) | 0.6 (3.1) | -0.5 (2.3)
  Cognitive function, Day 57: number analyzed (Participants) | 33 | 43 | 26 | 37
  Cognitive function, Day 57 | -0.3 (2.8) | -0.2 (2.8) | 0.2 (3.0) | -0.4 (2.6)
  Cognitive function, Day 85 | -0.2 (2.5) | 0.0 (3.1) | 0.7 (3.0) | -0.3 (3.0)
  Emotional, Day 29: number analyzed (Participants) | 35 | 44 | 28 | 37
  Emotional, Day 29 | 0.7 (4.4) | -1.1 (3.6) | -0.8 (4.2) | -0.3 (4.8)
  Emotional, Day 57: number analyzed (Participants) | 33 | 41 | 26 | 37
  Emotional, Day 57 | 0.7 (5.0) | -0.1 (4.6) | -0.1 (6.3) | -1.0 (5.1)
  Emotional, Day 85: number analyzed (Participants) | 38 | 47 | 40 | 37
  Emotional, Day 85 | 0.5 (4.6) | -0.6 (3.7) | -0.6 (5.8) | -1.3 (4.9)

33. Secondary Outcome: LTSE Phase: Change From Baseline in Quality of Life as Determined by PBC-40 Scale
Description: PBC-40 is a disease-specific quality of life questionnaire, which consists of 5 Domains(score ranges):general symptoms (score range 7-35), itch (3-15), fatigue (11-55), cognitive function (6-30) and emotional (1-15); higher scores indicated worse outcomes.The 40 questions from the PBC-40 questionnaire were scored from 1 (lowest impact of PBC on QoL) to 5 (representing highest impact); Higher scores indicate worse quality of life. Outcomes of 'never', 'not at all' or 'strongly agree' are scored with 1, 'always', 'very much' or 'strongly disagree' with 5, with following exceptions: For questions 34-39 outcomes were scored in reverse,i.e., 'strongly agree' with 5, and 'strongly disagree' with 1. If less than 50% of the questions per domain were not answered, missing values were imputed by mean of the available question scores for that domain.If for any item multiple answers are given, most severe was used. Baseline = Day 85. Change from Baseline=post Baseline minus Baseline value.
Time Frame: Baseline and at 6 and 12 months
Population: Safety Population (N=78). Only those participants with data available at specified time points has been presented (n=66).
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | LTSE OCA Total
Number analyzed (Participants) | 66
Scores on a scale
  General symptoms, 6 months | 0.3 (3.0)
  General symptoms, 12 months: number analyzed (Participants) | 60
  General symptoms, 12 months | 0.3 (2.7)
  Itch, 6 months | 1.2 (3.6)
  Itch, 12 months: number analyzed (Participants) | 60
  Itch, 12 months | 0.5 (3.3)
  Fatigue, 6 months | -1.1 (5.1)
  Fatigue, 12 months: number analyzed (Participants) | 60
  Fatigue, 12 months | -1.7 (5.4)
  Cognitive function, 6 months | 0.1 (3.0)
  Cognitive function, 12 months: number analyzed (Participants) | 60
  Cognitive function, 12 months | -0.4 (3.3)
  Emotional, 6 months | -0.4 (4.4)
  Emotional, 12 months: number analyzed (Participants) | 60
  Emotional, 12 months | -1.0 (5.4)

34. Secondary Outcome: Double-blind Phase: Change From Baseline in Quality of Life as Determined by 5-Dimension (5-D) Domain Scale
Description: 5-D questionnaire has 5 domains: Duration, degree, direction, disability, distribution, and total score. Single item domain scores (duration, degree, direction)=range:1-5.Disability domain has 4 items=assess impact of itching on daily activities: sleep, leisure/social activities, housework/errands, work/school;score calculated as highest score on any of 4 items; disability domain range=1-5.For distribution domain only section "Mark whether itching has been present in following parts of your body over the last 2 weeks" was used. Number of affected body parts('present') is tallied(potential sum 0-16);sum was sorted into 5 scoring bins: sum 0-2= score 1,sum 3-5=score 2,sum 6-10=score 3, sum 11-13=score 4,sum 14-16=score 5. Distribution score range reported=1-5. For all domains, higher scores=worse outcomes. Total 5D score=summing domain scores; ranges:5(no pruritus) to25 (most severe pruritus); Higher scores=worse outcomes. Baseline=Day 0.Change from Baseline=post Baseline minus Baseline
Time Frame: Baseline and at Days 29, 57 and 85
Population: ITT Population (N=165). Only those participants with data available at specified time points has been presented (n=163).
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Obeticholic Acid (OCA) 10 Milligrams (mg) | OCA 25 mg | OCA 50 mg | Placebo
Number analyzed (Participants) | 38 | 47 | 40 | 38
Scores on a scale
  Total score, Day 29: number analyzed (Participants) | 35 | 42 | 25 | 35
  Total score, Day 29 | 2.6 (3.4) | 3.0 (4.7) | 4.4 (5.4) | -0.7 (2.9)
  Total score, Day 57: number analyzed (Participants) | 30 | 40 | 24 | 35
  Total score, Day 57 | 1.8 (4.5) | 2.6 (3.9) | 2.9 (3.3) | -1.8 (3.0)
  Total score, Day 85: number analyzed (Participants) | 37 | 43 | 36 | 36
  Total score, Day 85 | 1.3 (3.8) | 1.7 (4.0) | 4.2 (5.1) | -1.5 (3.8)
  Duration, Day 29: number analyzed (Participants) | 35 | 43 | 26 | 36
  Duration, Day 29 | 0.3 (0.9) | 0.7 (1.5) | 1.2 (1.6) | 0.1 (1.0)
  Duration, Day 57: number analyzed (Participants) | 32 | 41 | 25 | 35
  Duration, Day 57 | 0.4 (1.3) | 0.6 (1.1) | 0.5 (1.0) | -0.3 (0.7)
  Duration, Day 85: number analyzed (Participants) | 37 | 45 | 39 | 36
  Duration, Day 85 | 0.2 (0.8) | 0.4 (1.1) | 0.8 (1.2) | -0.2 (0.8)
  Degree, Day 29: number analyzed (Participants) | 35 | 44 | 26 | 36
  Degree, Day 29 | 0.5 (0.8) | 0.6 (1.0) | 1.0 (1.1) | 0.0 (0.6)
  Degree, Day 57: number analyzed (Participants) | 32 | 43 | 25 | 36
  Degree, Day 57 | 0.3 (1.0) | 0.7 (1.0) | 0.7 (1.0) | -0.2 (0.8)
  Degree, Day 85: number analyzed (Participants) | 37 | 45 | 39 | 37
  Degree, Day 85 | 0.4 (0.9) | 0.6 (1.0) | 0.9 (1.1) | -0.2 (0.7)
  Direction, Day 29: number analyzed (Participants) | 35 | 44 | 25 | 35
  Direction, Day 29 | 0.5 (1.1) | 0.2 (1.5) | -0.2 (1.6) | -0.3 (1.2)
  Direction, Day 57: number analyzed (Participants) | 30 | 43 | 24 | 36
  Direction, Day 57 | 0.0 (1.3) | 0.1 (1.5) | -0.2 (1.4) | -0.7 (1.4)
  Direction, Day 85: number analyzed (Participants) | 37 | 46 | 36 | 36
  Direction, Day 85 | -0.2 (1.5) | -0.2 (1.5) | 0.1 (1.4) | -0.5 (1.5)
  Disability, Day 29: number analyzed (Participants) | 35 | 43 | 27 | 36
  Disability, Day 29 | 0.7 (1.2) | 0.7 (1.2) | 1.3 (1.5) | -0.3 (0.9)
  Disability, Day 57: number analyzed (Participants) | 32 | 42 | 26 | 36
  Disability, Day 57 | 0.4 (1.1) | 0.6 (1.1) | 0.8 (1.2) | -0.4 (1.1)
  Disability, Day 85: number analyzed (Participants) | 38 | 45 | 40 | 37
  Disability, Day 85 | 0.3 (1.2) | 0.6 (1.2) | 1.0 (1.4) | -0.4 (1.2)
  Distribution, Day 29: number analyzed (Participants) | 35 | 44 | 28 | 37
  Distribution, Day 29 | 0.6 (0.9) | 0.8 (1.5) | 1.4 (1.6) | -0.2 (0.9)
  Distribution, Day 57: number analyzed (Participants) | 33 | 43 | 26 | 37
  Distribution, Day 57 | 0.5 (1.1) | 0.8 (1.2) | 1.4 (1.3) | -0.2 (0.8)
  Distribution, Day 85 | 0.6 (0.9) | 0.8 (1.2) | 1.2 (1.5) | -0.2 (1.0)

35. Secondary Outcome: Double-blind Phase: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant administered a medicinal product without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. TEAEs were defined as any AE that started or worsened in severity on or after the first dose of study treatment.
Time Frame: Up to Day 85
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Obeticholic Acid (OCA) 10 Milligrams (mg) | OCA 25 mg | OCA 50 mg | Placebo
Number analyzed (Participants) | 38 | 48 | 41 | 38
Participants
  Any TEAE | 34 | 47 | 41 | 32
  Any SAE | 0 | 1 | 5 | 1

36. Secondary Outcome: Double-blind Phase: Change From Baseline in Pruritus Visual Analog Scale (VAS)
Description: A VAS questionnaire was used to assess participant's pruritus. The pruritus VAS measures participant's perception of itch on a continuous scale with score ranged from 0 = no itching and 10 = worst possible itching; higher score indicates worse outcomes. Baseline was defined as the last observed value before the first dose of investigational product (Day 0). Change from Baseline was defined as value of post Baseline minus Baseline value.
Time Frame: Baseline and at Days 29, 57 and 85
Population: ITT Population (N=165). Only those participants with data available at specified time points has been presented (n=152).
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Obeticholic Acid (OCA) 10 Milligrams (mg) | OCA 25 mg | OCA 50 mg | Placebo
Number analyzed (Participants) | 36 | 41 | 40 | 35
Scores on a scale
  Day 29: number analyzed (Participants) | 35 | 40 | 26 | 32
  Day 29 | 11.5 (19.5) | 17.8 (26.3) | 22.8 (33.2) | -2.6 (16.3)
  Day 57: number analyzed (Participants) | 31 | 39 | 24 | 33
  Day 57 | 7.0 (25.7) | 15.4 (24.7) | 13.7 (25.7) | -10.7 (19.6)
  Day 85 | 6.5 (22.2) | 12.9 (24.5) | 17.2 (28.9) | -5.8 (20.5)

37. Secondary Outcome: LTSE Phase: Number of Participants With TEAEs and SAEs
Description: An AE was any untoward medical occurrence in a participant administered a medicinal product without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. TEAEs were defined as any AE that started or worsened in severity on or after the first dose of study treatment.
Time Frame: Up to 12 Months
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | LTSE OCA Total
Number analyzed (Participants) | 78
Participants
  Any TEAE | 76
  Any SAE | 5

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected Up to Day 85 for Double-blind phase and up to 12 Months for LTSE phase.
Description: AEs and SAEs were collected in Safety Population that comprised of all randomized participants who received at least 1 dose of investigational product.
Groups:
- LTSE OCA Total: Participants from the double-blind phase entered the open-label LTSE phase of the study. A total of 7 participants entered the LTSE within 2 weeks of completing the double-blind phase. Participants initially started dosing at less than or equal to (<=) 10 mg daily OCA and continued daily dosing at >10 mg to ≤25 mg OCA. Entry of 71 participants from double-blind phase to LTSE phase was delayed up to 10 months due to administrative reasons.
Arm/Group | Obeticholic Acid (OCA) 10 Milligrams (mg) | OCA 25 mg | OCA 50 mg | Placebo | LTSE OCA Total
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/48 | 0/41 | 0/38 | 0/78
Serious Adverse Events (participants affected / at risk) | 0/38 | 1/48 | 5/41 | 1/38 | 5/78
Other Adverse Events (participants affected / at risk) | 34/38 | 47/48 | 41/41 | 32/38 | 76/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Obeticholic Acid (OCA) 10 Milligrams (mg) (N=38) | OCA 25 mg (N=48) | OCA 50 mg (N=41) | Placebo (N=38) | LTSE OCA Total (N=78)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Biliary cirrhosis primary (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystocele (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Obeticholic Acid (OCA) 10 Milligrams (mg) (N=38) | OCA 25 mg (N=48) | OCA 50 mg (N=41) | Placebo (N=38) | LTSE OCA Total (N=78)
Pruritus (Skin and subcutaneous tissue disorders) | 18 (23) | 41 (52) | 33 (60) | 19 (21) | 68
Dry Eye (Eye disorders) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 0
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0) | 4 (4) | 1 (1) | 6
Constipation (General disorders) | 3 (3) | 4 (4) | 3 (4) | 3 (3) | 7
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 4 (4) | 3 (4) | 3 (3) | 4
Nausea (Gastrointestinal disorders) | 4 (4) | 3 (3) | 4 (4) | 1 (1) | 4
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0
Fatigue (General disorders) | 7 (8) | 3 (3) | 5 (7) | 5 (6) | 10
Pyrexia (General disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 4 (4) | 0 (0) | 5
Headache (Nervous system disorders) | 3 (3) | 5 (7) | 7 (8) | 4 (6) | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0
Oopharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 0 (0) | 1 (1) | 0
Oedema Peripheral (General disorders) | 0 | 0 (0) | 0 (0) | 0 (0) | 5
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 10
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 10
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All publications or lectures involving study material or data will be submitted for approval to Intercept Pharmaceuticals prior to submission to any journal/publication/lecture according to the clinical trial agreement.